CLINICAL TRIAL: NCT01089855
Title: Phase IV Open Non Comparative Trial to Evaluate Efficacy and Safety of Tegretol® in Diabetes Neuropathy Pain.
Brief Title: Efficacy and Tolerability of Carbamazepine CR in Diabetic Neuropathy Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTEG111ZMA01
Record Dates: First submitted 2010-03-17; First posted 2010-03-19 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2011-02

CONDITIONS: Neuropathic Pain
Keywords: Neuropathic Pain; Brief Pain Inventory; DN4 questionnaire; ElectroCardioGram
MeSH Terms: conditions — Neuralgia | interventions — Carbamazepine

ARMS (1):
- Carbamazepine (Experimental)
  Interventions: Drug: Carbamazepine

INTERVENTIONS:
Drug: Carbamazepine

SUMMARY:
The trial is designed to evaluate the efficacy and tolerability of carbamazepine in neuropathic pain in diabetic patients

ELIGIBILITY:
Inclusion Criteria:

* Diabetes patients with Diabetes neuropathy DN4 > or equal to 4
* Male or female aged from 21 to 65 years
* Informed consent
* HbA1C < 11%

Exclusion Criteria:

* Prior Hospitalization for Acido- cetosis
* Prior hospitalization for severe hypoglycemia
* Pregnancy
* Hepatitis
* Diabetes foot
* AVB (auriculo-ventricular conduction disturbance)
* Patient treated by antidepressant drugs
* Patient treated with other antiepileptic drug
* Patients with blood ion disturbance
* Patient with neutropenia
* Glaucoma
* Bladder Adenoma
* Alcohol abuse
* Creatinin clearance < 60 ml/ minute

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2009-12; Primary Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
The decrease of neuropathic pain in diabetic patients using Brief Pain Inventory scale (BPI) | 12 weeks

SECONDARY OUTCOMES:
Evaluate the tolerability of carbamazepine (including Adverse Events, Serious Adverse Events and abnormal laboratory finding) | 12 weeks
Evaluate the quality of life | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigational Site, Rabat, Morocco